CLINICAL TRIAL: NCT02346448
Title: Endoscopic Sphincterotomy vs. Balloon Dilation for Assessment of Pancreatitis: A Prospective Randomized Multicenter Trial
Brief Title: Endoscopic Sphincterotomy vs. Balloon Dilation for Assessment of Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helios Albert-Schweitzer-Klinik Northeim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HELIOS 4/8/14
Record Dates: First submitted 2015-01-20; First posted 2015-01-27 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Pancreatitis
Keywords: endoscopic sphincterotomy; balloon dilation; adverse events; pancreatitis; bleeding
MeSH Terms: conditions — Pancreatitis; Hemorrhage | interventions — Sphincterotomy, Endoscopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- endoscopic sphincterotomy (Active Comparator): performing endoscopic sphincterotomy of papilla of Vater during ERCP Device: standard sphincterotome
  Interventions: Procedure: endoscopic sphincterotomy
- balloon dilatation for 3 minutes (Active Comparator): Balloon dilatation of papilla of Vater for 3 minutes during ERCP using 10mm balloon Device: standard dilation balloon catheter (10mm size)
  Interventions: Procedure: balloon dilatation for 3 minutes
- balloon dilatation for 6 minutes (Active Comparator): Balloon dilatation of papilla of Vater for 6 minutes during ERCP using 10mm balloon Device: standard dilation balloon catheter (10 mm size)
  Interventions: Procedure: balloon dilatation for 6 minutes

INTERVENTIONS:
Procedure: endoscopic sphincterotomy — sphincterotomy during ERCP
  Arms: endoscopic sphincterotomy
Procedure: balloon dilatation for 3 minutes — balloon dilatation during ERCP using 10mm balloon
  Arms: balloon dilatation for 3 minutes
Procedure: balloon dilatation for 6 minutes — balloon dilatation during ERCP using 10mm balloon
  Arms: balloon dilatation for 6 minutes

SUMMARY:
One of the major elements of successful endoscopic retrograde cholangiopancreatography ( ERCP) is the timely and uncomplicated cannulation of the common bile duct (CBD) . Various factors may adversely affect the cannulation procedure of the CBD leading to complications (acute pancreatitis after ERCP, perforation of the duodenum , bleeding ). Endoscopic sphincterotomy is frequently required for interventional procedures (eg stone extraction). During sphincterotomy, incision of the orifice of the papilla will be performed by using a sphincterotome. Complications due to sphincterotomy are known: Bleeding, increased rates of acute pancreatitis, small bowel perforation and scarring with consecutive stenosis of the papilla. As an alternative to sphincterotomy, balloon dilatation using balloon catheters can be performed. As a result, bleeding complications and scarring as late effects might be prevented. Current data is limited in terms of the risk of acute pancreatitis after ERCP when using a balloon catheter.

This study aims to evaluate the incidence of acute pancreatitis and other complications after ERCP. Balloon dilatation of the papilla will be prospectively compared with endoscopic sphincterotomy in a randomized multicenter setting.

ELIGIBILITY:
Inclusion Criteria:

* independent indication for ERCP
* age ≥ 18 years
* patient is able to understand informed consent

Exclusion Criteria:

* S/p sphincterotomy
* pancreatic or CBD-stent in situ
* pregnant patient
* known chronic pancreatitis
* acute pancreatitis prior to intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
acute pancreatitis | one to 10 days
  Definition of acute pancreatitis: Serum lipase or amylase obtained 2 to 6 hours following ERCP + onset of abdominal pain after ERCP persisting for 24h+ need for analgesia

SECONDARY OUTCOMES:
severity of pancreatitis using the Imrie score system (according to Imrie et al.) | one to 10 days
  assessment of severity by Imrie score: mild pancreatitis defined by Imrie score <3, severe pancreatitis if Imrie score >=3
endoscopic perforation | one to two days
  signs of perforation after ERCP, proven by CT scan or surgery
major bleeding | one to two days
  any bleeding events associated with ERCP. Drop of Hemoglobin of > 2g/dl and signs of bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, PDDr.med., Study Director — Helios Albert-Schweitzer-Hospital; Volker Ellenrieder, ProfDr.med., Study Director — University Medical Center Göttingen
Locations (3):
- Germany (3):
  - Department of Gastroenterology, University Medical Center, Göttingen, Lower Saxony
  - HELIOS Albert-Schweitzer Hospital Northeim, Northeim, Lower Saxony
  - HELIOS Klinikum Erfurt, Erfurt, Thuringia